CLINICAL TRIAL: NCT04361916
Title: Home Care for Patients With COVID-19: Active Monitoring in Two Italian Health Units (Casale Monferrato and Torino)
Acronym: Mon-Covid
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: interrupted early due to the drastic reduction in the number of cases
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Mon-Covid
Record Dates: First submitted 2020-04-14; First posted 2020-04-24 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-08

CONDITIONS: COVID-19
Keywords: COVID-19; oximetry; active monitoring; home care
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: single arm, open label trial on active home monitoring strategy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- home care with active monitoring (Experimental): home care with active monitoring conducted by health workers with daily visit to patients.
  Interventions: Other: home care monitoring

INTERVENTIONS:
Other: home care monitoring — home care active monitoring of patients with suspected of confirmed COVID-19

SUMMARY:
Starting an early home management and monitoring of patients with suspected or confirmed COVID-19 to ensure a rapid and adequate transfer to hospital care.

Assess the feasibility of home monitoring in a pilot study to possibly extend it to a larger scale.

DETAILED DESCRIPTION:
The study will include adult patients with suspected or confirmed COVID-19 for whom home care is considered appropriate.

Trained health workers will conduct home care monitoring of pulmonary performance using oximetry, Quick Walk Test and Single Breath Count.

Monitoring will be done daily until disappearance of symptoms or hospitalization which will be requested by health workers or study coordination board on the basis of the monitoring results (blood oxygen level SpO2< 90% OR SpO2> 90% with desaturation index of at least 5% at Quick Walk Test)

ELIGIBILITY:
Inclusion criteria:

adult patients with suspected or confirmed COVID-19 for whom home care is considered appropriate.

Exclusion criteria: physical, mental or temporary impairments that preclude the conduction of the test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
SpO2 at hospital entry | 24 hours
  Peripheral blood saturation measured on arrival to the hospital

SECONDARY OUTCOMES:
in-hospital mortality | 30 days
  death during hospitalization
need of intubation | 30 days
  need of intubation
Percentage of hospitalized patients among those with recommendation of hospitalization | 30 days
  To evaluate the feasibility of active monitoring, we will consider the percentage of patients who will be actually hospitalized within 24 hours after the recommendation of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Guido Bertolini, MD, Principal Investigator — Mario Negri Institute for Pharmacological Research
Locations (1):
- Asl Alessandria, Casale Monferrato, Alessandria, Italy

IPD SHARING:
Plan to Share IPD: Yes
data will be available from the study sponsor upon legitimate request
Supporting Information: Study Protocol